CLINICAL TRIAL: NCT02437955
Title: Evaluating the National Fortification Policy in Senegal Assessment of Iron Bio-availability in Mother and Child Pairs From Wheat Flour Fortified With Iron With and Without Phenolic Containing Beverages
Brief Title: Fe Absorption in Mother and Child Pairs From Wheat Fortified With Iron With and Without Phenolic Containing Beverages
Acronym: Fe_Senegal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Cheikh Anta Diop University, Senegal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: EK 2014-N-37
Record Dates: First submitted 2015-04-15; First posted 2015-05-08 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Anemia; Deficiency, Nutritional, With Poor Iron Absorption
MeSH Terms: conditions — Anemia | interventions — Tea; Water

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- FESO4+T (Experimental): Ferrous sulfate fortified bread with tea
  Interventions: Other: Ferrous sulfate fortified bread with tea
- FESO4+W (Experimental): Ferrous sulfate fortified bread with water
  Interventions: Other: ferrous sulfate fortified bread with water
- FeFu+T (Experimental): Ferrous fumarate fortified bread with tea
  Interventions: Other: Ferrous fumarate fortified bread with tea
- FeFu+W (Experimental): Ferrous fumarate fortified bread with water
  Interventions: Other: Ferrous fumarate fortified bread with water

INTERVENTIONS:
Other: Ferrous sulfate fortified bread with tea — Fasting subjects will be served a wheat roll fortified with labelled ferrous sulfate and stable isotopes
  Arms: FESO4+T
Other: ferrous sulfate fortified bread with water — Fasting subjects will be served a wheat roll fortified with labelled ferrous sulfate and stable isotopes
  Arms: FESO4+W
Other: Ferrous fumarate fortified bread with tea — Fasting subjects will be served a wheat roll fortified with labelled Fe Fumarate and stable isotopes
  Arms: FeFu+T
Other: Ferrous fumarate fortified bread with water — Fasting subjects will be served a wheat roll fortified with labelled Fe Fumarate and stable isotopes
  Arms: FeFu+W

SUMMARY:
In Senegal, iron deficiency affects 39% of and 82% of women and children between 12 and 50 months indicating that iron deficiency is a major health problem. The government of Senegal has implemented a flour fortification program including iron and folate. Iron is a difficult mineral to add to foods efficiently due to its organoleptic properties and typical low bioavailability in man. The aim of this study is to determine iron absorption from fortified wheat flour consumed with a phenolic containing beverage in women and child pairs. The fortificants used will be Ferrous Fumarate and Ferrous Sulfate, and the effect of absorption inhibitors on the bioavailability from iron compounds not readily bioavailable is poorly investigated.

The bioavailability of the different iron compounds will be determined using stable iron isotopes. Sixteen pairs of women and children (n=34, children between 3-6 years, women between 18-45y) will be selected for participation in the study. After a screening, each women and child will receive 4 test meals consisting of a bread roll fortified stable isotopes with and without the tisane beverage. The first two test meals will be consumed on consecutive days. Two weeks after the second test meal a blood sample will be taken from each women and child before the third meal administration. After the forth test meal administration, and again two weeks later, the last blood sampling will take place and the study will be conducted for the subjects (duration 30 days). The samples will be sent to Zurich on dry ice for analysis for the following parameters: isotopic composition, H pylori infection, B vitamin status, Vitamin A status. In all samples, hemoglobin and iron status as well as inflammation status (CRP) will be determined.

DETAILED DESCRIPTION:
In this study each subject will act as his own control and receive all interventions. Iron absorption data from the different test meals will be therefore compared assessing within and subject effects (main outcomes). Secondary outcomes will also investigate between subject effects and co variates of iron absorption.

ELIGIBILITY:
Inclusion Criteria

* Mother and child are willing to participate in the study jointly

Specific inclusions criteria for mothers

* Body weight < 65 kg
* 17 ≤ BMI ≤ 25 (kg/m2)
* Non anemic (Hb ≥ 11,0 g/dl)
* Generally healthy and no chronic illnesses
* Non pregnant
* Non lactating
* No blood donation in the last 4 months
* No consumption of vitamin and nutritional supplements during and 2 weeks prior the study start.

Inclusion criteria for children:

* Age 3-6 years
* Generally healthy and no chronic illnesses
* no consumption of vitamin and mineral supplements during and 2 weeks prior the study start

Ages: 3 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Iron absorption measured as iron incorporation of stable isotopic labels in red blood cells 14 days after administration | Up to 8 Months after study start
  The effect of the consumption of tea (phenolic containing beverages) will be assessed the two iron fortification compounds. The interaction between beverage and compound on iron absorption will be tested. The analysis will be separately conducted for mothers and children.

SECONDARY OUTCOMES:
Correlation between iron absorption in mother and child pairs | Up to 8 Months after study start
  The correlation of iron absorption from the different test meals between in mother and child pairs will be assessed. A variable will be defined which will consist of the difference in iron absorption between each mother and child, within one mother child pair cluster. Determinants of this variable will be explored by linear regression, such as iron status, parity, age, gender, anthropometry, iron status, vitamin status (A, B2, B12, folate) h. pylori test and hepcidin.

CONTACTS AND LOCATIONS:
Overall Officials: Ndeye Fatou Ndiaye, PhD, Principal Investigator — Université Cheikh Anta Diop de Dakar, Sengal
Locations (1):
- Université Cheikh Anta Diop, Dakar, Senegal